CLINICAL TRIAL: NCT06156163
Title: Effectiveness of Perturbation Training in Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Tuğba Akgüller, lecturer, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: takguller
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
Keywords: low back pain; nonspecific low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perturbation Group (Experimental): Exercise program with progressive perturbation conditions
  Interventions: Other: Perturbation training
- Exercise Group (Active Comparator): Exercise program
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Perturbation training — The exercise program will be applied 2 days/week for 8 weeks, with the addition of progressive perturbation conditions.
  Arms: Perturbation Group
Other: Exercise — The exercise program will be applied 2 days/week for 8 weeks.
  Arms: Exercise Group

SUMMARY:
Nonspecific low back pain is defined as low back pain that cannot be associated with a specific identified pathology. Many methods such as patient education, medical treatment, physical modalities, exercise, manual therapy, massage, traction and cognitive behavioral therapy are used in the treatment of nonspecific low back pain. Spinal stabilization exercises, which are among the therapeutic exercises, aim to improve and improve muscle control to compensate for any loss of muscle movement caused by degenerative changes or injury. Perturbation training, which is among the neuromuscular exercises, is an intervention that aims to improve the control of rapid balance reactions and involves repetitive postural distortions. In perturbation training, the surface is moved in multiple directions with different forces and moments. The aim of this exercise is to develop the stabilization response that will be created by stresses applied from different directions. It is believed that the number of motor units participating in contraction and proprioceptive input will increase with perturbation exercise. Although the number of studies on low back pain is quite limited, it has been stated that applications that provide perturbation can reduce the incidence of low back pain and provide improvement in neuromuscular control of spinal stability. In the light of these data, the aim of this study is to investigate the effects of perturbation training given in addition to the exercise program on trunk muscle endurance, pain, disability, functionality, fear avoidance beliefs and quality of life parameters in individuals with nonspecific low back pain.

DETAILED DESCRIPTION:
Nonspecific low back pain is defined as low back pain that cannot be associated with a specific identified pathology. Many methods such as patient education, medical treatment, physical modalities, exercise, manual therapy, massage, traction and cognitive behavioral therapy are used in the treatment of nonspecific low back pain. In current guidelines, it has been reported that patient education and therapeutic exercises are treatment methods with a high level of evidence. Spinal stabilization exercises, which are among the therapeutic exercises, aim to improve and improve muscle control to compensate for any loss of muscle movement caused by degenerative changes or injury. With stabilization exercises, deep muscles are activated while excessive activity of superficial muscles is reduced. Thus, correcting muscle abnormalities and ensuring the correct function of the muscles supports the spine. Perturbation training, which is among the neuromuscular exercises, is an intervention that aims to improve the control of rapid balance reactions and involves repetitive postural distortions. In perturbation training, the surface is moved in multiple directions with different forces and moments. The aim of this exercise is to develop the stabilization response that will be created by stresses applied from different directions. It is believed that the number of motor units participating in contraction and proprioceptive input will increase with perturbation exercise. Previous studies have shown that the effects of perturbation training were mostly investigated in geriatric and neurological patient groups. However, current studies show that perturbation training is also applied to some orthopedic problems such as anterior cruciate ligament injury, shoulder pain, ankle instability and makes positive contributions to the healing process.

Although the number of studies on low back pain is quite limited, it has been stated that applications that provide perturbation can reduce the incidence of low back pain and provide improvement in neuromuscular control of spinal stability. In the light of these data, the aim of this study is to investigate the effects of perturbation training given in addition to the exercise program on trunk muscle endurance, pain, disability, functionality, fear avoidance beliefs and quality of life parameters in individuals with nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific low back pain persisting for at least 3 months
* Pain intensity at least 3 on VAS
* Ability to perceive verbal and written Turkish instructions
* Having signed the voluntary consent form

Exclusion Criteria:

* History of spinal surgery/trauma
* Low back cpain associated with other pathologies (Rheumatic diseases, malignancy, MS)
* Having herniation at the level of sequestration and extrusion
* Instability conditions such as spondylolysis and spondylolisthesis
* Use of painkillers and antidepressants
* Pregnancy
* Obesity (BMI≥30kg/m²)
* Orthopedic problems and chronic diseases that may prevent exercises
* FTR/steroid injection application within the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-12-16 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Trunk extensor endurance test | At baseline and after 8 weeks of intervention
  Individuals are asked to hang their trunks from the bed starting from the spina iliaca anterior superior and cross both arms on the shoulders. The legs are fixed by the practitioner over the gastrocnemius muscle. The test is started when the individuals maintain the horizontal position and the time they maintain the position is recorded in seconds.
Trunk flexor endurance test | At baseline and after 8 weeks of intervention
  The participant is positioned by the tester with the knees and hips at 90 degrees, the body at 60 degrees, the hands in a crossed position on both shoulders, and the soles of the feet firmly on the ground. The time this position can be maintained is recorded in seconds.
Bilater side bridge endurance test | At baseline and after 8 weeks of intervention
  For the left lateral plank test, the participants' feet are placed on top of each other, the right arm is perpendicular to the ground, the elbow is on the mat, the left arm is at chest level, and the left hand is on the right shoulder. When the individual is ready, he is asked to lift his hips with support from his elbows and feet. As soon as the test position is taken in which the shoulders, hips and feet are in the same direction, the time is started by the researcher. The period ends when the individual cannot maintain the position and body swings forward and backward.

SECONDARY OUTCOMES:
Pain intensity | At baseline and after 8 weeks of intervention
  The pain felt by the participants at rest, during activity and at night will be questioned with the "0-10 cm" Visual Analogue Scale (VAS). On VAS, 0 means "no pain" and 10 means "worst pain ever felt".
Disability | At baseline and after 8 weeks of intervention
  The disability levels of the participants will be evaluated with the 'Oswestry Disability Index (ODS)'. The survey contains 10 questions on 10 topics with 6 options. The increase in the total score is proportional to the increase in activity limitation.
Timed Up and Go Test | At baseline and after 8 weeks of intervention
  The 3-meter area in front of the chair is determined. The patient is asked to get up from the chair, walk this distance and sit down again. The elapsed time gives the result of the test and the time is recorded in seconds. The test is performed twice with a 1-minute interval and the average time is taken.
The Fear-Avoidance Beliefs Questionnaire (FABQ) | At baseline and after 8 weeks of intervention
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability.
  The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. [2] There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24).
Health-related quality-of-life | At baseline and after 8 weeks of intervention
  Individuals' health-related quality of life will be evaluated with Short Form-12/SF-12. With SF-12, two subscores are obtained: physical component summary (PBS) and mental component summary (MBS). While the FBÖ-12 score is obtained from the sub-dimensions of general health, physical functionality, physical role and body pain, the MBÖ-12 score is obtained from the social functionality, emotional role, mental health and energy sub-dimensions. Both FBÖ-12 and MBÖ-12 scores range from 0 to 100, with a higher score representing better health.
Patient Satisfaction | After 8 weeks of intervention
  Patient satisfaction with the treatment will be evaluated with the Global Rating of Change scale. Participants will be asked to rate their condition compared to baseline after an 8-week intervention period, indicating whether they had significantly improved, slightly improved, remained unchanged, slightly deteriorated, or significantly worsened in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Fitzgerald GK, Axe MJ, Snyder-Mackler L. The efficacy of perturbation training in nonoperative anterior cruciate ligament rehabilitation programs for physical active individuals. Phys Ther. 2000 Feb;80(2):128-40. PMID 10654060
- [Background] Schinkel-Ivy A, Huntley AH, Aqui A, Mansfield A. Does Perturbation-Based Balance Training Improve Control of Reactive Stepping in Individuals with Chronic Stroke? J Stroke Cerebrovasc Dis. 2019 Apr;28(4):935-943. doi: 10.1016/j.jstrokecerebrovasdis.2018.12.011. Epub 2019 Jan 7. PMID 30630753
- [Background] Schafer R, Schafer H, Platen P. Perturbation-based trunk stabilization training in elite rowers: A pilot study. PLoS One. 2022 May 19;17(5):e0268699. doi: 10.1371/journal.pone.0268699. eCollection 2022. PMID 35587490
- [Background] Arampatzis A, Schroll A, Catala MM, Laube G, Schuler S, Dreinhofer K. A random-perturbation therapy in chronic non-specific low-back pain patients: a randomised controlled trial. Eur J Appl Physiol. 2017 Dec;117(12):2547-2560. doi: 10.1007/s00421-017-3742-6. Epub 2017 Oct 19. PMID 29052033
- [Background] Evans K, Refshauge KM, Adams R. Trunk muscle endurance tests: reliability, and gender differences in athletes. J Sci Med Sport. 2007 Dec;10(6):447-55. doi: 10.1016/j.jsams.2006.09.003. Epub 2006 Dec 1. PMID 17141568
- [Background] Shamsi MB, Rezaei M, Zamanlou M, Sadeghi M, Pourahmadi MR. Does core stability exercise improve lumbopelvic stability (through endurance tests) more than general exercise in chronic low back pain? A quasi-randomized controlled trial. Physiother Theory Pract. 2016;32(3):171-8. doi: 10.3109/09593985.2015.1117550. Epub 2016 Feb 11. PMID 26864057